CLINICAL TRIAL: NCT05610501
Title: Ultrasound-guided Tru-Cut Biopsy in Pelvic Masses.
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: UZ Leuven, Leuven, Belgium (Unknown); Policlinico Universitario A. Gemelli, IRCSS, Rome, Italy. (Unknown); Charles University, Czech Republic (Other); Karolinska Institutet and Department of Obstetrics and Gynecology, Södersjukhuset, Stockholm, Sweden. (Unknown)
Responsible Party: Sponsor
Other Study IDs: S64793
Record Dates: First submitted 2022-09-28; First posted 2022-11-09 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Pelvic Cancer; Ovarian Cancer; Cervical Cancer; Uterus Cancer; Endometrial Cancer; Ovarian Neoplasms; Ovarian Carcinoma; Sarcoma Uterus; Metastatic Cancer
Keywords: Tru-cut; Ultrasound; Pelvic mass; Ovarian cancer; Gynaecologic oncology
MeSH Terms: conditions — Pelvic Neoplasms; Ovarian Neoplasms; Uterine Cervical Neoplasms; Uterine Neoplasms; Endometrial Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient population: All consecutive patients (> 18 years) undergoing a tru-cut biopsy at the participating centers during the study periof will be eligible for inclusion in the study.
  All biopsies will be performed by trained operators in gynecologic ultrasound and tru-cut biopsies. Tissue samples will be assessed by experienced pathologists, dedicated in gynecologic oncology. Data will be collected by reviewing patients' electronic medical file including data concerning further treatment-strategy and pathology reports. Patients' level of pain and overall experience will be assessed by an independent investigator not present during biopsy. This will be performed from 0-72h after the biopsy using a numeric rating scale (0-100). Safety and complication-rate will be assessed by both using the collected data and via postprocedural assessment and by phone after six weeks. Inclusion and exclusion criteria can be found elsewhere.
  Interventions: Procedure: Ultrasound guided tru-cut biopsy

INTERVENTIONS:
Procedure: Ultrasound guided tru-cut biopsy — Tru-cut biopsies can collect tissue specimens via a needle of 18G A tru-cut biopsy can be performed under the guidance of different imaging modalities including ultrasound

SUMMARY:
In a transvaginal tru-cut biopsy, guided by ultrasound, a needle is inserted through the vaginal wall into a pelvic lesion and a few pieces of tissue are obtained for examination.

This clinical trial is organized to evaluate the safety and efficacy of transvaginal tru-cut biopsy in a large group of patients with tumors in the small pelvis.

DETAILED DESCRIPTION:
Ovarian cancer is known to be the 4th most lethal tumour in women and has the highest mortality rate of all gynaecological malignancies. In most women, the disease is not diagnosed until advanced stage [1]. Moreover, the pelvis and ovaries in particular, are also a common place for secondary metastases. In 4% of ovarian masses, metastasis can be found from a tumour with another primary origin [2]. In primary ovarian cancer, patients may benefit from either primary debulking surgery or neoadjuvant therapy, depending on tumour staging and patients' comorbidities [5]. In recurrent disease treatment may include surgery, radiotherapy or systemic therapy, depending on primary tumour histology, extent of recurrence, previous treatment and disease-free interval [6-8]. In pelvic masses with ultrasound features suggesting metastatic disease, management will be guided by the origin of the primary tumour [9,10]. Therefore, histological diagnosis is important to select the optimal treatment strategy.

Tissue sampling by diagnostic laparoscopy or explorative laparotomy requires general anaesthesia and hospital admission, leading to higher costs and to potential surgical morbidity. Moreover, diagnostic laparoscopy is associated with a risk of port-site metastasis, ranging from 0.3-0.4% in endometrial and cervical cancer [11] and even 17-49% in advanced ovarian cancer [12,13].

Minimally invasive procedures for diagnosis include fine-needle aspiration and tru-cut biopsy.

At fine-needle aspiration the quantity and integrity of the tissue is limited, enabling cytological evaluation only [14]. Tru-cut biopsy results in a higher specificity compared to fine needle biopsy and it enables histological examination including immunohistochemistry [15,16].

A tru-cut biopsy can be performed under the guidance of different imaging modalities including ultrasound, Computed Tomography (CT) and Magnetic Resonance Imaging (MRI). However, percutaneous CT-guided biopsies of deep pelvic masses are challenging because vital structures often obstruct the needle pathway [17].

Previous studies have investigated the use of ultrasound-guided biopsies for the assessment of abdominal and pelvic masses which showed a high diagnostic adequacy and minimal complication rate [4,16,18-25]. This can be done by percutaneous transabdominal approach , a transvaginal or transrectal approach.

The main goal of this prospective study is to evaluate the safety and tissue yield of ultrasound guided transvaginal or transrectal tru-cut biopsy in patients with pelvic tumors. Secondly, factors affecting the reliability of the biopsy-results will be analyzed, as well as patients' experience and pain. Finally, a comparison of biopsy results and final histological diagnosis will be performed in those patients undergoing surgical management.

5. Study aims Primary Aim The main goal of our study is 1) to evaluate the safety (defined as absence of procedure-related complications) and 2) tissue yield (defined as sufficient amount of tissue for histological analysis) of ultrasound guided transvaginal or transrectal tru-cut biopsy in patients with pelvic masses.

Secondary Aims

* Analyzing factors affecting the safety and tissue yield. (The influence of selected variables such as number of biopsies per target lesion, length of the shot (15 vs 22 mm), thickness of needle (16-18 G), target lesion, target lesion size, histotypes etc. on these outcomes will be assessed.)
* Assessment of patients' overall experience, assessment of pain and discomfort during the procedure and afterwards.
* Comparison of biopsy result with final histological diagnosis: histological type (only in patients finally undergoing surgery)

Study design Prospective multicentric observational study

ELIGIBILITY:
Inclusion Criteria:

* 1. Following lesion criteria applicable for biopsy:

  1. Lesion safely accessible (no visceral or vessel interposition; in the case of a transvaginal approach no vaginal stenosis (severe atrophy - virgo - vaginismus); within reach of biopsy needle)
  2. Solid component present (purely cystic lesions excluded)

     2. Biopsy for research purposes, the following is applicable: Patients with a gynecological tumor eligible for participation in academic or commercial clinical trials requesting a biopsy for translational research. For the current study, which is observational, we do not intend to take additional biopsies outside routine clinical practice, but only biopsies requested for participation in other (interventional) studies on systemic treatment in gynecologic oncology.

     3. In case of a diagnostic biopsy, one of the following inclusion criteria should be applicable:

  <!-- -->

  1. Suspicious primary disseminated gynecologic tumor (tumor itself or metastasis) Patients with a presumable new diagnosis of a disseminated pelvic tumor where histological confirmation of disease is necessary before the possibility to start a specific oncologic treatment and

     * Are invalid candidates for primary (radical) surgery due to comorbidities or poor overall general wellbeing
     * Are invalid candidates for primary (radical) surgery due to the extensive disease-spread according to imaging and/or diagnostic laparoscopy
  2. Suspicious primary disseminated NON-gynecologic tumor (tumor itself or metastasis)
  3. Patients with possible recurrence of a gynecological tumor (cervix, myometrial, endometrial, ovarian etc), where histological confirmation of disease recurrence is necessary before the possibility to start a surgical or systemic intervention.
  4. Patients with possible recurrence of a presumably non-gynecological tumor, where histological confirmation of disease recurrence is necessary before start of treatment.
  5. Solitary tumor of unknown histology localized in vaginal wall, parametria, retroperitoneum or uterine wall and can be punctured without spilling in abdominal cavity.

Exclusion Criteria:

- 1. Patients < 18 years 2. Clotting defect or anticoagulation therapy, precluding a safe biopsy even with adapted therapy regimen.

3. Vaginal or pelvic infection 4. Poor performance status contraindicating any specific oncologic treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients (> 18 years) undergoing a tru-cut biopsy at the collaborating centers for a pelvic mass.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Safety | 6 weeks
  Defined as absence of procedure-related complications. Procedure related complications will be graded by Clavien-Dindo classification.
Tissue yield | 6 weeks after procedure
  Defined as sufficient amount of tissue for histological analysis. This will be a binary variable based on the pathology report.

SECONDARY OUTCOMES:
Factor 1 affecting safety and tissue yield | 6 weeks
  A number of biopsies per target lesion,
Factor 2 affecting safety and tissue yield | 6 weeks
  The length of the needle shot (15 vs 22 mm).
Factor 3 affecting safety and tissue yield | 6 weeks
  The thickness of needle (16-18 Gauge).
Factor 4 affecting safety and tissue yield | 6 weeks
  The target lesion histotype - categorical variable defined by the tumour type.
Factor 5 affecting safety and tissue yield | 6 weeks
  The target lesion size in mm.
Patient experience | 3 days
  Assessment of patients' overall experience using VAS-Score.
Patient pain score | 3 days
  Assessment of patients' pain and discomfort during the procedure using VAS-Score.
Histological diagnosis | 6 weeks
  Comparison of biopsy result with final histological diagnosis: histological type (only in patients finally undergoing surgery). Binary variable indicating agreement.

CONTACTS AND LOCATIONS:
Locations (4):
- UZ Leuven, Leuven, Belgium
- First Faculty of Medicine, Charles University, Prague, Czechia
- Fondazione Policlinico Universitario A. Gemelli, IRCSS, Rome, Italy
- Department of Clinical Science and Education, Karolinska Institutet and Department of Obstetrics and Gynecology, Södersjukhuset, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chandra A, Pius C, Nabeel M, Nair M, Vishwanatha JK, Ahmad S, Basha R. Ovarian cancer: Current status and strategies for improving therapeutic outcomes. Cancer Med. 2019 Nov;8(16):7018-7031. doi: 10.1002/cam4.2560. Epub 2019 Sep 27. PMID 31560828
- [Background] Van Calster B, Van Hoorde K, Valentin L, Testa AC, Fischerova D, Van Holsbeke C, Savelli L, Franchi D, Epstein E, Kaijser J, Van Belle V, Czekierdowski A, Guerriero S, Fruscio R, Lanzani C, Scala F, Bourne T, Timmerman D; International Ovarian Tumour Analysis Group. Evaluating the risk of ovarian cancer before surgery using the ADNEX model to differentiate between benign, borderline, early and advanced stage invasive, and secondary metastatic tumours: prospective multicentre diagnostic study. BMJ. 2014 Oct 15;349:g5920. doi: 10.1136/bmj.g5920. PMID 25320247
- [Background] Testa AC, Ferrandina G, Timmerman D, Savelli L, Ludovisi M, Van Holsbeke C, Malaggese M, Scambia G, Valentin L. Imaging in gynecological disease (1): ultrasound features of metastases in the ovaries differ depending on the origin of the primary tumor. Ultrasound Obstet Gynecol. 2007 May;29(5):505-11. doi: 10.1002/uog.4020. PMID 17444565
- [Background] Epstein E, Van Calster B, Timmerman D, Nikman S. Subjective ultrasound assessment, the ADNEX model and ultrasound-guided tru-cut biopsy to differentiate disseminated primary ovarian cancer from metastatic non-ovarian cancer. Ultrasound Obstet Gynecol. 2016 Jan;47(1):110-6. doi: 10.1002/uog.14892. PMID 25925783
- [Background] Vergote I, Trope CG, Amant F, Kristensen GB, Ehlen T, Johnson N, Verheijen RH, van der Burg ME, Lacave AJ, Panici PB, Kenter GG, Casado A, Mendiola C, Coens C, Verleye L, Stuart GC, Pecorelli S, Reed NS; European Organization for Research and Treatment of Cancer-Gynaecological Cancer Group; NCIC Clinical Trials Group. Neoadjuvant chemotherapy or primary surgery in stage IIIC or IV ovarian cancer. N Engl J Med. 2010 Sep 2;363(10):943-53. doi: 10.1056/NEJMoa0908806. PMID 20818904
- [Background] Peiretti M, Zapardiel I, Zanagnolo V, Landoni F, Morrow CP, Maggioni A. Management of recurrent cervical cancer: a review of the literature. Surg Oncol. 2012 Jun;21(2):e59-66. doi: 10.1016/j.suronc.2011.12.008. Epub 2012 Jan 14. PMID 22244884
- [Background] Al Rawahi T, Lopes AD, Bristow RE, Bryant A, Elattar A, Chattopadhyay S, Galaal K. Surgical cytoreduction for recurrent epithelial ovarian cancer. Cochrane Database Syst Rev. 2013 Feb 28;2013(2):CD008765. doi: 10.1002/14651858.CD008765.pub3. PMID 23450588
- [Background] Bradford LS, Rauh-Hain JA, Schorge J, Birrer MJ, Dizon DS. Advances in the management of recurrent endometrial cancer. Am J Clin Oncol. 2015 Apr;38(2):206-12. doi: 10.1097/COC.0b013e31829a2974. PMID 23764681
- [Background] Van Calster B, Van Hoorde K, Froyman W, Kaijser J, Wynants L, Landolfo C, Anthoulakis C, Vergote I, Bourne T, Timmerman D. Practical guidance for applying the ADNEX model from the IOTA group to discriminate between different subtypes of adnexal tumors. Facts Views Vis Obgyn. 2015;7(1):32-41. PMID 25897370
- [Background] Agnes A, Biondi A, Ricci R, Gallotta V, D'Ugo D, Persiani R. Krukenberg tumors: Seed, route and soil. Surg Oncol. 2017 Dec;26(4):438-445. doi: 10.1016/j.suronc.2017.09.001. Epub 2017 Sep 12. PMID 29113663
- [Background] Martinez A, Querleu D, Leblanc E, Narducci F, Ferron G. Low incidence of port-site metastases after laparoscopic staging of uterine cancer. Gynecol Oncol. 2010 Aug 1;118(2):145-50. doi: 10.1016/j.ygyno.2010.03.011. Epub 2010 May 7. PMID 20451983
- [Background] Vergote I, Marquette S, Amant F, Berteloot P, Neven P. Port-site metastases after open laparoscopy: a study in 173 patients with advanced ovarian carcinoma. Int J Gynecol Cancer. 2005 Sep-Oct;15(5):776-9. doi: 10.1111/j.1525-1438.2005.00135.x. PMID 16174223
- [Background] Heitz F, Ognjenovic D, Harter P, Kommoss S, Ewald-Riegler N, Haberstroh M, Gomez R, Barinoff J, Traut A, du Bois A. Abdominal wall metastases in patients with ovarian cancer after laparoscopic surgery: incidence, risk factors, and complications. Int J Gynecol Cancer. 2010 Jan;20(1):41-6. doi: 10.1111/IGC.0b013e3181c443ba. PMID 20057285
- [Background] Malmstrom H. Fine-needle aspiration cytology versus core biopsies in the evaluation of recurrent gynecologic malignancies. Gynecol Oncol. 1997 Apr;65(1):69-73. doi: 10.1006/gyno.1996.4606. PMID 9103393
- [Background] Chojniak R, Isberner RK, Viana LM, Yu LS, Aita AA, Soares FA. Computed tomography guided needle biopsy: experience from 1,300 procedures. Sao Paulo Med J. 2006 Jan 5;124(1):10-4. doi: 10.1590/s1516-31802006000100003. Epub 2006 Apr 3. PMID 16612456
- [Background] Fischerova D, Cibula D, Dundr P, Zikan M, Calda P, Freitag P, Slama J. Ultrasound-guided tru-cut biopsy in the management of advanced abdomino-pelvic tumors. Int J Gynecol Cancer. 2008 Jul-Aug;18(4):833-7. doi: 10.1111/j.1525-1438.2007.01015.x. Epub 2007 Aug 30. PMID 17764453
- [Background] Gupta S, Nguyen HL, Morello FA Jr, Ahrar K, Wallace MJ, Madoff DC, Murthy R, Hicks ME. Various approaches for CT-guided percutaneous biopsy of deep pelvic lesions: anatomic and technical considerations. Radiographics. 2004 Jan-Feb;24(1):175-89. doi: 10.1148/rg.241035063. PMID 14730045
- [Background] Volpi E, Zola P, De Grandis T, Rumore A, Volpe T, Sismondi P. Transvaginal sonography in the diagnosis of pelvic malignant recurrence: integration of sonography and needle-guided biopsy. Ultrasound Obstet Gynecol. 1994 Mar 1;4(2):135-8. doi: 10.1046/j.1469-0705.1994.04020135.x. PMID 12797207
- [Background] Sheth SS, Angirish J. Transvaginal trucut biopsy in patients with abdominopelvic mass. Int J Gynaecol Obstet. 1995 Jul;50(1):27-31. doi: 10.1016/0020-7292(95)02433-d. PMID 7556856
- [Background] Faulkner RL, Mohiyiddeen L, McVey R, Kitchener HC. Transvaginal biopsy in the diagnosis of ovarian cancer. BJOG. 2005 Jul;112(7):991-3. doi: 10.1111/j.1471-0528.2005.00619.x. PMID 15958006
- [Background] Zikan M, Fischerova D, Pinkavova I, Dundr P, Cibula D. Ultrasound-guided tru-cut biopsy of abdominal and pelvic tumors in gynecology. Ultrasound Obstet Gynecol. 2010 Dec;36(6):767-72. doi: 10.1002/uog.8803. PMID 20737454
- [Background] Kong TW, Chang SJ, Paek J, Cho H, Lee Y, Lee EJ, Ryu HS. Transvaginal Sonography-Guided Core Biopsy of Adnexal Masses as a Useful Diagnostic Alternative Replacing Cytologic Examination or Laparoscopy in Advanced Ovarian Cancer Patients. Int J Gynecol Cancer. 2016 Jul;26(6):1041-7. doi: 10.1097/IGC.0000000000000728. PMID 27206281
- [Background] Park JJ, Kim CK, Park BK. Ultrasound-Guided Transvaginal Core Biopsy of Pelvic Masses: Feasibility, Safety, and Short-Term Follow-Up. AJR Am J Roentgenol. 2016 Apr;206(4):877-82. doi: 10.2214/AJR.15.15702. Epub 2016 Feb 25. PMID 26913556
- [Background] Zahedi R, Uppal S, Mendiratta-Lala M, Higgins EJ, Nettles AN, Maturen KE. Percutaneous image-guided pelvic procedures in women with gynecologic cancers: utilization, complications, and impact on patient management. Abdom Radiol (NY). 2016 Dec;41(12):2460-2465. doi: 10.1007/s00261-016-0882-9. PMID 27565659
- [Background] Lin SY, Xiong YH, Yun M, Liu LZ, Zheng W, Lin X, Pei XQ, Li AH. Transvaginal Ultrasound-Guided Core Needle Biopsy of Pelvic Masses. J Ultrasound Med. 2018 Feb;37(2):453-461. doi: 10.1002/jum.14356. Epub 2017 Sep 8. PMID 28885718